CLINICAL TRIAL: NCT03855007
Title: Prospective Clinical Study to Observe the Efficacy and Safety of Iguratimod in Rheumatoid Arthritis and Early Rheumatoid Arthritis Patients for 6 Months Treatment in China
Brief Title: The Clinical Efficacy and Safety of Iguratimod in RA and Early RA Patients for 6 Months Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Qiang Shu, Chief Physician, Qilu Hospital of Shandong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Iguratimod-ERA QiluH
Record Dates: First submitted 2019-02-15; First posted 2019-02-26 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Arthritis, Rheumatoid
Keywords: Iguratimod
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — iguratimod; T 614; Methotrexate; Hydroxychloroquine; prednylidene; Prednisone

STUDY DESIGN:
Intervention Model Description: Drug: Iguratimod（T-614），25mg, po, twice per day (Bid) prescribed at the beginning and adjusted due to patient response. Then may titer down until the endpoint.
  Drug: Methotrexate （MTX），7.5mg to 15mg, po, once per week (Qw) prescribed if needed and adjusted due to patient response or unacceptable toxicity develops.
  Drug: Hydroxychloroquine （HCQ），200mg, po, twice per day (Bid) prescribed if needed and adjusted due to patient response.
  Drug: Prednisone （Pred）： 5-15mg, po, once per day (Qd) prescribed if needed and adjusted due to patient response
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Iguratimod (Experimental): The participants plan to be treated with iguratimod alone, or along with methotrexate (MTX), hydroxychloroquine (HCQ) , prednisone (Pred) step by step
  Interventions: Drug: Iguratimod; Drug: MTX; Drug: HCQ; Drug: Pred

INTERVENTIONS:
Drug: Iguratimod — Iguratimod tablet，25mg, po, twice per day (Bid) prescribed at the beginning and adjusted due to patient response. Then may titer down until the endpoint.
  Other Names: T-614
Drug: MTX — MTX，7.5mg to 15mg, po, once per week (Qw) prescribed if needed and adjusted due to patient response or unacceptable toxicity develops.
  Other Names: methotrexate
Drug: HCQ — HCQ，200mg, po, twice per day (Bid) prescribed if needed and adjusted due to patient response.
  Other Names: Hydroxychloroquine
Drug: Pred — Pred, 5-15mg, po, once per day (Qd) prescribed if needed and adjusted due to patient response
  Other Names: Prednisone

SUMMARY:
This study is designed to observed prospectively the efficacy and safety of 6 months treatment of iguratimod alone, or with methotrexate (MTX), hydroxychloroquine (HCQ) and prednisone step by step on Chinese rheumatoid arthritis (RA) and early rheumatoid arthritis (ERA) patients who were naïve or shown insufficiency response or intolerance to DMARDs. If volunteered, patients who completed the 6-month study can continue to follow our plans for 24 months.

DETAILED DESCRIPTION:
This study will enroll 200 cases of rheumatoid arthritis (RA) and early rheumatoid arthritis (ERA) patients in China, who are naïve or shown insufficiency response or intolerance to DMARDs. The participants plan to be treated with iguratimod alone, or along with methotrexate (MTX)/ hydroxychloroquine (HCQ) / prednisone (Pred) step by step for 6 months if participants are in medium or high disease activity (DAS28≥3.2). Participants can choose to continue the study up to 24 months.The efficacy and safety of 6 months and 24 months Iguratimod treatment in RA and ERA patients will be evaluated with DAS28-ESR and other disease activity indices.

ELIGIBILITY:
Inclusion Criteria: -

1. RA: Patients diagnosed based on 1987 ACR classification criteria for rheumatoid arthritis(RA);
2. ERA: Subjects diagnosed by the 2010 American College of Rheumatology/European League Against Rheumatism (ACR/EULAR); or by 2012 Chinese classification criteria of early rheumatoid arthritis (ERA), and not match the 1987 ACR criteria for RA.
3. Age ≥16 years;
4. Extra-articular manifestations (such as pulmonary fibrosis, proteinuria, leukopenia and peripheral neuropathy ) of RA patients are stable or no significant progress;
5. Patients can be naïve to any DMARDs, or relapse due to DMARDs drug suspended;
6. Patients have a history of using csDMARDs including csDMARDs（methotrexate，leflunomide, hydroxychloroquine, sulfasalazine, tacrolimus) , any biologic DMARDs（TNFi，tocilizumab or Tofacitinib），glucocorticoid (prednisone，methylprednisolone) or Chinese traditional Medicine（including tripterygium Glycosides, sinomenine）for 3 months, but couldn't achieve clinical remission or intolerance；

Exclusion Criteria:

1. Patients with acute or chronic infections such as active bacterial, viral, fungal, tuberculosis infection or active hepatitis B;
2. Platelet counts(PLT) <80 x 10^9 / L, or white blood cell (WBC) <3 x 10^9 / L;
3. Propionate acid aminotransferase (ALT) or aspartate aminotransferase (AST) is two times higher than the upper limit of normal;
4. Renal insufficiency: serum Cr ≥ 176 umol / L;
5. Pregnant or nursing women (breastfeeding) ；
6. Patients has a history of malignancy (cure time in less than 5 years);
7. Patients with severe or poorly controlled hypertension, diabetes or cardiac dysfunction;
8. Other comorbidities that cannot be treated with immune suppressants. In addition, once patients experience severe adverse drug reactions、ineffective treatment or rapid progression of rheumatoid arthritis, then quit this research.

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
The percentage of patients who achieve clinical remission at week 24 using European League Against Rheumatism (EULAR) response criteria DAS28 | week 24
  The percentage of patients whose Disease Activity Score in 28 Joints (DAS28) achieve remission（DAS28-ESR≤ 2.6）and Low Disease Activity (DAS28-ESR ≤ 3.2). The DAS28 is a composite score derived from 4 of these measures，that is the count of tender joint count（TJC, 0-28）and swollen joint count（SJC, 0-28）, measure erythrocyte sedimentation rate (ESR, mm/h) or C reactive protein (CRP, mg/L) and to make a patient assessment of disease activity i.e. 'global assessment of health' (GH) using a 100 mm visual analogue scale (VAS) with 0 = best, 100 = worst. DAS28 values were calculated as follows: DAS28- ESR = 0.56√(TJC) + 0.28√(SJC) + 0.70 ln ESR + 0.014 x GH. High disease activity: DAS28-ESR > 5.1; Moderate disease activity: 5.1≥ DAS28 > 3.2 to 5.1; Low disease activity (LDA) and Remission mean Clinical remission.

SECONDARY OUTCOMES:
The percentage of patients who achieve clinical remission using DAS28-ESR at week 12 | week 12
  The percentage of patients whose DAS28 achieve remission（DAS28-ESR≤ 2.6）and Low Disease Activity (DAS28-ESR ≤ 3.2) at week 12.
The percentage of patients who achieve clinical remission using DAS28-ESR at week 48 | week 48
  The percentage of patients whose DAS28 achieve remission（DAS28-ESR≤ 2.6）and Low Disease Activity (DAS28-ESR ≤ 3.2) at week 12.response states were classified as follows: good responders were patients with an improvement from baseline (△DAS28-ESR) of > 1.2 and a DAS28-ESR at week 12 ≤ 3.2. Moderate responders: △DAS28 > 1.2 and still DAS28 > 3.2 at week 12, or 1.2 ≥△DAS28 > 0.6 and DAS28 ≤ 5.1 at week 12. Nonresponders：△DAS28 ≤0.6 or DAS28 >5.1 at week 12. DAS28-defined remission was classified as a score of <2.6.
The percentage of patients who achieve clinical remission using DAS28-ESR at week 96 | week 96
  The percentage of patients whose DAS28 achieve remission（DAS28-ESR≤ 2.6）and Low Disease Activity (DAS28-ESR ≤ 3.2) at week 12Nonresponders：△DAS28 ≤0.6，or DAS28 >5.1 at week 24. DAS28-defined remission was classified as a score of <2.6.
Percentage of Disease Activity Score 28 (DAS28) -ESR Criteria Responders at week 12 | week 12
  △DAS28 indicates the decline of DAS28-ESR from the baseline to week 12. EULAR response states were classified as follows: good responders were patients with an improvement from baseline (△DAS28-ESR) of > 1.2 and a DAS28-ESR at week 12 ≤ 3.2. Moderate responders: △DAS28 > 1.2 and still DAS28 > 3.2 at week 12, or 1.2 ≥△DAS28 > 0.6 and DAS28 ≤ 5.1 at week 12. Nonresponders：△DAS28 ≤0.6 or DAS28 >5.1 at week 12. DAS28-defined remission was classified as a score of <2.6.
Percentage of Disease Activity Score 28 (DAS28)-ESR Criteria Responders at week 24 | week 24
  EULAR response states were classified as follows: DAS28-ESR Good responders: △DAS28 > 1.2 and DAS28 ≤3.2 at week 24. Moderate responders：△DAS28 > 1.2 and still DAS28 > 3.2 at week 24; or 1.2 ≥△DAS28 > 0.6 and DAS28 ≤ 5.1 at week 24. Nonresponders：△DAS28 ≤0.6，or DAS28 >5.1 at week 24. DAS28-defined remission was classified as a score of <2.6.
Percentage of Disease Activity Score 28 (DAS28)-ESR Criteria Responders at week 48 | week 48
  EULAR response states were classified as follows: DAS28-ESR Good responders: △DAS28 > 1.2 and DAS28 ≤3.2 at week 24. Moderate responders：△DAS28 > 1.2 and still DAS28 > 3.2 at week 24; or 1.2 ≥△DAS28 > 0.6 and DAS28 ≤ 5.1 at week 24. Nonresponders：△DAS28 ≤0.6，or DAS28 >5.1 at week 24. DAS28-defined remission was classified as a score of <2.6.
Percentage of Disease Activity Score 28 (DAS28)-ESR Criteria Responders at week 96 | week 96
  EULAR response states were classified as follows: DAS28-ESR Good responders: △DAS28 > 1.2 and DAS28 ≤3.2 at week 24. Moderate responders：△DAS28 > 1.2 and still DAS28 > 3.2 at week 24; or 1.2 ≥△DAS28 > 0.6 and DAS28 ≤ 5.1 at week 24. Nonresponders：△DAS28 ≤0.6，or DAS28 >5.1 at week 24. DAS28-defined remission was classified as a score of <2.6.
Percentage of participants achieving ACR/EULAR remission at week 12 | week 12
  If all of the following 4 parameters are fulfilled, it is defined as remission: TJC ≤ 1, SJC ≤ 1, CRP ≤ 1 mg/dL, Patient global assessment（PGA） ≤ 1 cm (on a visual analog scale ranging from 0-10 cm, with higher scores indicating severe disease).
Percentage of participants achieving ACR/EULAR remission at week 24 | week 24
  If all of the following 4 parameters are fulfilled, it is defined as remission: TJC ≤ 1, SJC ≤ 1, CRP ≤ 1 mg/dL, Patient global assessment（PGA） ≤ 1 cm (on a visual analog scale ranging from 0-10 cm, with higher scores indicating severe disease).
Percentage of participants achieving ACR/EULAR remission at week 48 | week 48
  If all of the following 4 parameters are fulfilled, it is defined as remission: TJC ≤ 1, SJC ≤ 1, CRP ≤ 1 mg/dL, Patient global assessment（PGA） ≤ 1 cm (on a visual analog scale ranging from 0-10 cm, with higher scores indicating severe disease).
Percentage of participants achieving ACR/EULAR remission at week 96 | week 96
  If all of the following 4 parameters are fulfilled, it is defined as remission: TJC ≤ 1, SJC ≤ 1, CRP ≤ 1 mg/dL, Patient global assessment（PGA） ≤ 1 cm (on a visual analog scale ranging from 0-10 cm, with higher scores indicating severe disease).
Percentage of American College of Rheumatology [ACR] 20 Criteria Responders every 3 months | Up to week 96
  Percentage of American College of Rheumatology [ACR] 20 Criteria Responders every 3 months
Change from baseline Simplified Disease Activity Index (SDAI) | Up to week 96
  The SDAI is a composite score derived from these measures，that is the count of tender joint count（TJC, 0-28）, swollen joint count（SJC, 0-28）, C-reactive protein (CRP, mg/L), Patient global assessment（PGA）and physician global assessment（PHGA）, each of the last two was assessed on a visual analog scale ranging from 0-10 cm, with higher scores indicating severe disease. SDAI score will be calculated with formula SDAI = TJC + SJC + PGA+PHGA+ CRP. SDAI score exceeding 26 is considered high disease activity; 11 <SDAI ≤26，moderate disease activity; 3.3 <SDAI ≤11, low disease activity; remission is SDAI score ≤ 3.3.
Change from baseline Clinical Disease Activity Index (CDAI) | Up to week 96
  CDAI is a composite score derived from these measures，that is the count of tender joint count（TJC, 0-28）, swollen joint count（SJC, 0-28）, Patient global assessment（PGA）and physician global assessment（PHGA）, each of the last two was CDAI score will be calculated with formula CDAI = TJC + SJC + PGA + PHGA. CDAI > 22 is considered high disease activity; 10 <CDAI ≤ 22, moderate disease activity; 2.8 <CDAI ≤10, low disease activity; remission is CDAI score ≤2.8.
Change From Baseline in C-reactive Protein (CRP) | Up to week 96
  Change from Baseline in C-reactive Protein (CRP), a component index of ACR20 and SDAI, CRP will be measured with blood samples.
Change From Baseline in Erythrocyte Sedimentation Rate (ESR) | Up to week 96
  Change from Baseline in ESR, that is a component index of ACR20, DAS28-ESR and SDAI, ESR will be measured with blood samples.
Change from baseline Health Assessment Questionnaire Disability Index (HAQ-DI) | Up to week 96
  Change from Baseline in HAQ-DI, a participant assessed measure of health assessment, shaveing eight dimensions of functional activity: pruning, dressing, rising, eating, walking, personal hygiene, reach, grip, and other routine activities. Each item on a single scale has 4 degrees ranging from 0 (no functional difficulty) to 3 (unable to do), with higher scores indicating severe disease.
Incidence of participant withdrawal | Up to week 96
  Percentage of participants who withdraw from this study.
Number of participants with"adverse events (AEs)" | Up to week 96
  An AE is any untoward medical occurrence in a subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Number of participants with"adverse events (AEs)"i.e. physical exam abnormalities，vital sign abnormalities，laboratory value abnormalities，symptom or disease (new or exacerbated) temporally associated with the use of a medicinal product.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Lv, Dr., Study Director — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No